CLINICAL TRIAL: NCT04699084
Title: The Evaluation of Mozart Music on Pain and Respiratory Rate After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prolepsis Institute for Preventive, Environmental and Occupational Medicine (Other)
Responsible Party: Principal Investigator, Dimitrios Linos, Principal Investigator, Prolepsis Institute for Preventive, Environmental and Occupational Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUTHYROID
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants were assigned to two groups. One group underwent a music intervention postoperatively, while the other received only usual postoperative care (control group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Patients received music intervention and usual postoperative care.
  Interventions: Other: Mozart music
- Control Group (No Intervention): Patients received only postoperative usual care.

INTERVENTIONS:
Other: Mozart music — A 20-minute piece composed by W.A Mozart ( Sonata K. 448 in D Major for 2 pianos) was applied in music group, directly after the arrival of patients in the Post Anesthesia Care Unit (PACU), while they were receiving usual postoperative care.
  Arms: Music Group

SUMMARY:
To investigate the effect of Mozart music on postoperative pain and physiological parameters in patients after total thyroidectomy.

DETAILED DESCRIPTION:
Postoperative pain is a major concern in postsurgical patients. Meanwhile, there is a general consensus on minimizing the use of analgesic drugs in patients undergoing total thyroidectomy. Therefore, alternative methods need to be investigated in order to reduce postoperative pain. Although the clinical importance of music has been recognised in other pathological situations, further research is needed to investigate the effect of music on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for total thyroidectomy under general anesthesia

Exclusion Criteria:

* Visual impairments
* Hearing impairments
* Severe anxiety or other psychiatric disorders
* History of chronic pain
* Past complications during anesthesia or surgery
* American Society of Anesthesiologists (ASA) physical status beyond II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Change of VAS was evaluated; from the beginning (time of arrival at the PACU, baseline), to the middle (10 minutes after surgery), to the end of the music intervention (20 minutes after surgery) at the PACU and to 2 hours after surgery in the ward.
  Postoperative Pain was measured with the Visual Analogue Scale (VAS). This is a straight horizontal line of fixed length, usually 100 mm. The ends of the line are defined as the extreme limits of the measured parameter (pain). Specifically, the left end signifies the complete absence of pain and the right end represents the worst possible pain. Patients were asked to rate their pain by indicating a point on the straight line. Higher VAS scores mean more pain intensity. The more is the reduction of VAS score from the baseline measurement, the better is the outcome.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Change of blood pressure was evaluated during the first postoperative day.
  Blood pressure was measured by a patient's monitor.
Heart rate | Change of heart rate was evaluated during the first postoperative day.
  Heart rate was measured by a patient's monitor.
Respiratory rate | Change of respiratory rate was evaluated during the first postoperative day.
  Respiratory rate was measured by a care provider.
Oxygen saturation | Change of oxygen saturation was evaluated during the first postoperative day.
  Oxygen saturation was measured by a patient's monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Linos, MD, Ph.D., Principal Investigator — Hygeia Hospital, National and Kapodistrian University of Athens
Locations (1):
- Hygeia Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tripyla N, Katsas K, Karagkouni K, Liosis I, Ntelis S, Linos D. Evaluation of the effect of Mozart music on pain and respiratory rate after thyroidectomy. Hormones (Athens). 2023 Mar;22(1):113-119. doi: 10.1007/s42000-022-00421-7. Epub 2022 Nov 22. PMID 36418659